CLINICAL TRIAL: NCT03231696
Title: Visibility - A Novel Classification Score of Sono-visibility of Anatomical Structures in Peripheral Nerve Blocks
Brief Title: Visibility - Classification of Sono-visibility of Anatomical Structures in Peripheral Nerve Blocks
Acronym: Visibility
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jurgen Birnbaum, Senior physician of the Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK, Charite University, Berlin, Germany
Other Study IDs: Visibility
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Anesthesia, Local; Anesthesia
Keywords: nerve block; peripheral nerve stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving Regional Anesthesia: All patients 18 years or older with a peripheral nerve block at Charité - Universitätsmedizin Berlin Campus Charite Mitte from 2012 to 2016.

SUMMARY:
We assessed the visibility of peripheral nerves while ultrasound guided blockades with a novel scoring system to evaluate differences in visibility of different nerves.

DETAILED DESCRIPTION:
We assessed the visibility of peripheral nerves while ultrasound guided blockades with a novel scoring system to evaluate differences in visibility of different nerves.

VIS(visibility) 1 easy identification and instant visualisation of all structures VIS 2 identification and visualisation of all structures after some corrections VIS 3 identification and visualisation of structures only unsure VIS 4 identification and visualisation of all structures impossible VIS 5 no structures seen. We amended a sub-project in which assessed the visibility in protective nerve stimulated nerve blocks in 46 patients.

ELIGIBILITY:
Inclusion Criteria (study sample N=1200):

* peripheral nerve block by ultrasound guidance
* age ≥ 18 years

Exclusion Criteria:

* contraindications for regional anesthesia

Inclusion Criteria (study sample as of amendment n=46):

* peripheral nerve block by ultrasound guidance
* age ≥ 18 years

Exclusion Criteria:

* contraindications for regional anesthesia (study sample n=46)
* using not the standard ultrasound machine
* performing not a standard regional anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years or older with a peripheral nerve block at Charité - Universitätsmedizin Berlin Campus Charite Mitte from 2012 to 2016.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visibility | During regional block (an average of 1 hour)
  The ultrasound visibility of the nerve scored by a 5-step scale.

SECONDARY OUTCOMES:
Additional analgesia | During surgery (an average of 4 hours)
  The need and amount of additional analgetic drugs while the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Birnbaum, MD, Principal Investigator — Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No